CLINICAL TRIAL: NCT06557694
Title: Effect of COVID-19 Infection on Obstertric Complications and Maternal Outcomes
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Nabil Ageez, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR750/7/24
Record Dates: First submitted 2024-08-15; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Infection; Obstetric Complication; Maternal Outcomes
MeSH Terms: conditions — COVID-19; Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection: Data collected included maternal demographics, medication during pregnancy, the gestational week when COVID-19 was diagnosed, antenatal diseases occurring after COVID-19 detection during pregnancy, intrauterine growth retardation (IUGR), small for gestational age (SGA), fetal distress, intrauterine fetal demise (IUFD), intrapartum complications, gestational age (GA) at delivery, mode of delivery, postpartum hemorrhage (PPH), admission to the maternal ICU, birth weight, admission to the NICU, and the indication for NICU hospitalization
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collected included maternal demographics, medication during pregnancy, the gestational week when COVID-19 was diagnosed, antenatal diseases occurring after COVID-19 detection during pregnancy, intrauterine growth retardation (IUGR), small for gestational age (SGA), fetal distress, intrauterine fetal demise (IUFD), intrapartum complications, gestational age (GA) at delivery, mode of delivery, postpartum hemorrhage (PPH), admission to the maternal ICU, birth weight, admission to the NICU, and the indication for NICU hospitalization Pregnancy outcomes included mode of delivery, gestational age at delivery, pre-eclampsia, and postpartum hemorrhage (defined as an estimated blood loss of 1,000 mL or greater).

SUMMARY:
This study aimed to evaluate the effect of COVID-19 infection on obstetric complications and maternal outcomes.

DETAILED DESCRIPTION:
During the SARS-CoV-2 pandemic, pregnant women were reported to have a higher susceptibility to COVID-19 infection. Pregnant women who tested positive for SARS-CoV-2 are at higher risk of a severe form of COVID-19, associated with higher rates of intensive care unit (ICU) admission and increased needs for respiratory support, compared to the age-matched non-pregnant population.

Women infected during pregnancy also have an increased risk of adverse pregnancy outcomes including preterm-birth, with a significant proportion secondary to iatrogenic preterm birth due to maternal illness. Infection with SARS-CoV-2 during pregnancy has also been reported to be associated with a higher risk of stillbirth directly or indirectly caused by the virus.

Infected pregnant patients tended to present asymptomatically with pre-Delta and Omicron variants, and symptomatically with Delta variant. A previous systematic review suggested that people who are pregnant did not have an increased risk of SARS-CoV-2 infection or symptomatic COVID-19, but they were at risk of severe COVID-19 compared with those who were not pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* Pregnant women with COVID-19 infection diagnosed either by PCR or rapid test.

Exclusion Criteria:

• Patients vaccinated for COVID-19 before or during the current pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: This retrospective study was carried out on 260 pregnant women with COVID-19 infection who presented in Tanta University Hospitals in the period from January 2021 to December 2022 with approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy related complications | For one month
  Pregnancy related complications as preterm birth, preeclampsia, intrauterine fetal demise (IUFD), increased cesarean section rate, postpartum hemorrhagic gastroenteritis (HGE) were collected

SECONDARY OUTCOMES:
Intensive care unit admission rate | For one month
  Intensive care unit admission rate was collected.
Use of mechanical ventilation | For one year
  Use of mechanical ventilation was collected.
Incidence of death | For one month
  Incidence of death was collected.
Apgar score | For 5 minutes post-intervention
  Apgar score is a quick test performed on a baby at 1 and 5 minutes after birth. The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.